CLINICAL TRIAL: NCT06049147
Title: Randomized, Double Blind, Placebo Controlled "First-in-human" Study to Assess the Safety and Tolerability of Single Ascending Oral Doses and Multiple Oral Doses of MBF-015 in Healthy Young Volunteers
Brief Title: Study to Assess the Safety and Tolerability of MBF-015 in Healthy Young Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medibiofarma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MBF-015CT-01; 2020-005318-16 (EudraCT Number)
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Safety and Pharmacokinetic
Keywords: Histone deacetylase inhibitor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- MBF-015 4mg oral single dose (Experimental): Drug: MBF-015 oral single dose. MBF-015 4 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 4 mg oral capsule
- MBF-015 8 mg oral single dose (Experimental): Drug: MBF-015 oral single dose. Two 4 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 4 mg oral capsule
- MBF-015 16 mg oral single dose (Experimental): Drug: MBF-015 oral single dose. One 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- MBF-015 32 mg oral single dose (Experimental): Drug: MBF-015 oral single dose. Two 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- MBF-015 64 mg oral single dose (Experimental): Drug: MBF-015 oral single dose. Four 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- MBF-015 8 mg oral multiple dose (Experimental): Drug: MBF-015 oral single daily dose during five days. Two 4 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 4 mg oral capsule
- MBF-015 16 mg oral multiple dose (Experimental): Drug: MBF-015 oral single daily dose during five days. One 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- MBF-015 32 mg oral multiple dose (Experimental): Drug: MBF-015 oral single daily dose during five days. Two 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- MBF-015 64 mg oral multiple dose (Experimental): Drug: MBF-015 oral single daily dose during five days. Four 16 mg strength hard gelatin capsules
  Interventions: Drug: MBF-015 16 mg oral capsule
- Placebo single dose (Placebo Comparator): Placebo Hard gelatin capsules filled with cellulose microcrystalline. One single administration
  Interventions: Drug: Placebo
- Placebo multiple dose (Placebo Comparator): Placebo Hard gelatin capsules filled with cellulose microcrystalline. Single daily dose during five days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBF-015 4 mg oral capsule — MBF-015 oral capsules Histone deacetylase inhibitor
  Arms: MBF-015 4mg oral single dose; MBF-015 8 mg oral multiple dose; MBF-015 8 mg oral single dose
Drug: MBF-015 16 mg oral capsule — MBF-015 oral capsules Histone deacetylase inhibitor
  Arms: MBF-015 16 mg oral multiple dose; MBF-015 16 mg oral single dose; MBF-015 32 mg oral multiple dose; MBF-015 32 mg oral single dose; MBF-015 64 mg oral multiple dose; MBF-015 64 mg oral single dose
Drug: Placebo — Hard gelatin capsules filled with cellulose microcrystalline
  Arms: Placebo multiple dose; Placebo single dose

SUMMARY:
This is a single center, randomised, double blind, placebo controlled clinical study to assess the safety and tolerability of MBF-015 in healthy volunteers.This clinical phase I trial is divided in two stages and involves, first, a single ascending dose (SAD) study in healthy young male volunteers and then a multiple ascending dose (MAD) study in healthy young men and woman. MBF-118 is developed for the treatment of multiple sclerosis.

DETAILED DESCRIPTION:
This clinical phase I trial is divided in two stages. The first stage will be a dose escalation study without therapeutic benefit, in which MBF-015 will be administered as single oral ascending dose to healthy young male volunteers. Up to four different rising doses will be tested (4 mg, 8 mg, 16 mg, 32 mg, 64 mg) in groups/cohorts of 8 participants. Thus, five groups/cohorts will participate. For each dose level/group, the participants will be randomized to active or placebo with 2 participants being randomly assigned to placebo and 6 to the active drug. First, one volunteer will receive active drug and another one will receive placebo (subgroup 1); after at least 72h of safety and tolerability assessment a second subgroup of 3 volunteers will receive 2 active drug and 1 placebo; after at least another 72h of safety and tolerability parameters assessment, a third subgroup of 3 volunteers will receive the active drug. After evaluation of safety parameters of corresponding dose level, the process will replicate one week afterwards in the following dosages.

The second stage will be a dose escalation study without therapeutic benefit, in which MBF-015 will be administered as single oral daily dose, during 5 days to young male and female healthy volunteers. Up to four different rising dose levels will be tested (8 mg, 16 mg, 32 mg, and 64 mg) in cohorts of 8 subjects that are randomised to active treatment and placebo (6:2) and divided into three subsequent treatment blocks, as described above in the first stage.

The pharmacokinetics profile of MBF-015 will be also assessed at each dose level tested of the Single ascending dose study and the multiple ascending dose study. The 64 mg SAD part will also be used to measure the product concentration in cerebrospinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* To be included in the single dose study, subjects should meet all the following criteria at the screening visit:

  1. Healthy male subjects, 18-45 years (inclusive) of age at the time of enrolment.
  2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m)2.
  3. Normal clinical records and physical examination.
  4. Laboratory tests (haematology and biochemistry) within the range of normal values, according to the Biochemistry laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
  5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ Diastolic Blood Pressure (DBP) between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
  6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
  7. To be able to understand the nature of the study and comply with all their requirements.
  8. Free acceptance to participate in the study should be stated in an informed consent document signed by the volunteer which must be approved by the Clinical Research Ethic Committee (CREC).

For the multiple dose study in healthy male and female volunteers, subjects meeting all the following inclusion criteria at screening visit:

1. Healthy male and female subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination at screening and baseline.
4. Laboratory tests (haematology, biochemistry and urinalysis) within the range of normal values, according to the laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
7. To be able to understand the nature of the study and comply with all their requirements.
8. Free acceptance to participate in the study by obtains signed informed consent form approved by the CREC.
9. Females must be of non childbearing potential (i.e. surgically sterile) or have to use contraceptive measures ( non-hormonal) such as condom, diaphragm or cervical / vault caps with spermicide until 28 days post administration

Exclusion Criteria:

* For the single dose study and multiple dose study meeting any of the following criteria at screening visit will be excluded from entry into the study:

  1. History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 gr/day for men.
  2. Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day) and grape juice.
  3. Background of idiosyncrasy, food intolerance, hypersensitivity or adverse reactions to any drug or Galenic form.
  4. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
  5. Intake of any medication within 2 weeks prior taking the study treatment (except for use of paracetamol in short-term symptomatic treatments), including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), or any enzymatic inductor or inhibitor within 3 months before the drug administration.
  6. Positive serology for hepatitis B, C or HIV.
  7. Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, haematological, neurological disease or other chronic diseases.
  8. History of psychiatric diseases or epileptic seizures.
  9. 12 lead ECG obtained at screening with PR interval ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
  10. Having undergone major surgery during the previous 6 months.
  11. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc.) from 6 months prior to drug administration.
  12. Participation in other clinical trials during the previous 90 days (drug to drug period) in which an investigational drug or a commercially available drug was tested.
  13. Donation of blood during the 4 weeks preceding the drug administration.
  14. Severe or moderate acute illness 4 weeks before drug administration.
  15. Clinically significant abnormal laboratory values (as determined by the PI) at the screening evaluation.
  16. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract
  17. Positive results of the drugs at screening period or 24h before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the PI).
  18. Female with positive results from pregnancy test or breast-feeding (only in MAD stage)
  19. A positive Covid-19 diagnosis prior to admission to the hospital.
  20. A medical history of brain or spinal disease that would interfere with lumbar puncture, CSF circulation or safety assessment, including tumours or abnormalities by MRI or computed tomography (CT), subarachnoid hemorrhage, suggestion of raised intracranial pressure on MRI or ophthalmic examination, spinal stenosis or curvature, chiari malformation, hydrocephalus, syringomyelia, tethered spinal cord syndrome and connective tissue disorders such as Ehlers-Danlos syndrome and Marfan syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | Day 1 through Day 8
  Classification based in the Medical Dictionary for Regulatory Activities (MedDRa) Adverse Events will be qualified according to the definitions and values stated in CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Martinez, Principal Investigator — CIM-Sant Pau Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- CIM-Sant Pau Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No